CLINICAL TRIAL: NCT02910856
Title: Infective Endocarditis in the Elderly: Description of the Geriatric Characteristics and Their Influence on Therapeutic Care and the Morbidity and Mortality at 3 Months (ELDERL-IE)
Brief Title: Infective Endocarditis in the Elderly
Acronym: ELDERL-IE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Fondation Cœur et Recherche (Unknown)
Responsible Party: Principal Investigator, Christine Selton-Suty, Doctor, Central Hospital, Nancy, France
Other Study IDs: PSS 2014/ELDERL-IE-SELTON/SR
Record Dates: First submitted 2016-08-25; First posted 2016-09-22 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
ELDERL-IE is a multicenter national prospective observational study.

The main objective is to describe geriatric characteristics (comorbidities, cognitive status, autonomy, nutritional status, balance and walking) in patients aged 75 years or older with infective endocarditis (IE).

The secondary objectives are to assess the impact of geriatric features on the medico - surgical care and on morbidity and mortality at 3 months after the end of the hospitalization, and to describe the initial clinical presentation and diagnostic modalities in the IE elderly.

DETAILED DESCRIPTION:
Population monitoring:

Clinical, therapeutic, biological, microbiological, echocardiographic and geriatric data are collected. (M-2/3 before inclusion; D-15 before inclusion; D0; M3; vital status at 1 year)

ELIGIBILITY:
Inclusion Criteria :

* all patients older than 75 years are eligible if they are considered and treated as a case of IE by physicians ensuring their medical care.
* the patient should be treated in one of the clinical sites participating at the study.
* the patient should benefit during initial hospitalization of a geriatric assessment, in addition to the usual clinical and therapeutic management of such patients.

Exclusion criteria :

* patients not fulfilling the criteria of definite or possible endocarditis according to Duke modified by Li diagnostic classification that will be applied after collection of all the data at the discharge of the patient.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients older than 75 years are eligible if they are considered and treated as a case of IE by physicians ensuring their medical care.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline geriatric characteristics at 3 months | 3 months after inclusion
  OMS score

SECONDARY OUTCOMES:
Three months mortality | 3 months after inclusion
  Mortality rate at 3 months
One year mortality | 1 year after inclusion
  Mortality rate at 1 year
Change from baseline geriatric characteristics at 3 months | 3 months after inclusion
  Karnofsky'score
Change from baseline geriatric characteristics at 3 months | 3 months after inclusion
  Score MNA

CONTACTS AND LOCATIONS:
Overall Officials: Christine Selton-Suty, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Central Hospital - University Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Forestier E, Fraisse T, Roubaud-Baudron C, Selton-Suty C, Pagani L. Managing infective endocarditis in the elderly: new issues for an old disease. Clin Interv Aging. 2016 Sep 2;11:1199-206. doi: 10.2147/CIA.S101902. eCollection 2016. PMID 27621607
- [Result] Forestier E, Roubaud-Baudron C, Fraisse T, Patry C, Gavazzi G, Hoen B, Carauz-Paz P, Moheb-Khosravi B, Delahaye F, Sost G, Paccalin M, Nazeyrollas P, Strady C, Alla F, Selton-Suty C; AEPEI and the GInGer Elderl-IE study group; AEPEI and the GInGer Elderl-IE study group. Comprehensive geriatric assessment in older patients suffering from infective endocarditis. A prospective multicentric cohort study. Clin Microbiol Infect. 2019 Oct;25(10):1246-1252. doi: 10.1016/j.cmi.2019.04.021. Epub 2019 May 2. PMID 31055167
- [Result] Forestier E, Selton-Suty C, Roubaud-Baudron C. Managing infective endocarditis in older patients: do we need a geriatrician? Aging Clin Exp Res. 2021 Mar;33(3):719-722. doi: 10.1007/s40520-019-01400-6. Epub 2019 Nov 22. PMID 31758501
- [Result] N'cho-Mottoh MB, Erpelding ML, Roubaud C, Delahaye F, Fraisse T, Dijos M, Ennezat PV, Fluttaz A, Richard B, Beaufort C, Nazeyrollas P, Brasselet C, Pineau O, Tattevin P, Curlier E, Iung B, Forestier E, Selton-Suty C. The impact of transoesophageal echocardiography in elderly patients with infective endocarditis. Arch Cardiovasc Dis. 2023 May;116(5):258-264. doi: 10.1016/j.acvd.2023.04.001. Epub 2023 Apr 25. PMID 37147149